CLINICAL TRIAL: NCT04660461
Title: Response to Oral Lansoprazole of Inorganic Pyrophosphate Levels in Patients With Grönblad-Stranberg Disease (Pseudoxanthoma Elasticum)
Acronym: FIMPXE2016-01
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT 2016-004021-16; FIM-PXE-2016-01 (Other: FIMABIS)
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Grönblad-Stranberg Disease (Pseudoxanthoma Elasticum)
Keywords: Grönblad-Stranberg Disease; Pseudoxathoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum | interventions — Lansoprazole

STUDY DESIGN:
Intervention Model Description: Clinical trial, double blind, placebo controlled, randomized and crossed groups of patients in two stages, that receive a treatment with lansoprazole and placebo during 8 weeks with wash-ot period of 15 days
Who Masked: Participant, Investigator
Masking Description: The masking of the drug to produce the cecum will be carried out by the Pharmacy on University Hospital Virgen de la Macarena accredited by the AEMPS. The medication for this clinical trial will be prepared by the Pharmacy on University Hospital Virgen de la Macarena in Seville ; the lansoprazole capsules and their placebo will be re-encapsulated in larger ones to maintain the cecum. The proposed doses used are those used in mild/moderate gastro-oesophageal diseases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Randomized placebo-controlled, parallel-group study, crossover-design (Experimental)
  Interventions: Drug: Lansoprazole 30mg; Drug: Placebo
- 2. Randomized placebo-controlled, parallel-group study, crossover-design (Experimental)
  Interventions: Drug: Lansoprazole 30mg; Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole 30mg — Subjects are randomized to recieve Lansoprazole 30mg/day or placebo during 8 weeks. After a washing-out period of 15 days, subjects will receive the other treatment (cross-over design) during 8 weeks
Drug: Placebo — Subjects are randomized to recieve Lansoprazole 30mg/day or placebo during 8 weeks. After a washing-out period of 15 days, subjects will receive the other treatment (cross-over design) during 8 weeks

SUMMARY:
Protocol code and version: FIM-PXE-2016-01 Version 1.4

Trial title: "Response to oral lansoprazole of inorganic pyrophosphate levels in patients with Grönblad- Stranberg disease (Pseudoxanthoma Elasticum)"

Trial design: Double-blind, placebo-controlled, randomised, two-stage crossover clinical trial, with each patient serving as their own control and reducing the number of patients to confirm our hypothesis.

Principal Investigator: Dr. Pedro Valdivielso Felices Participating centres Virgen de la Victoria's Universitary Hospital in Malaga and Virgen de la Macarena's Universitary Hospital in Seville.

Duration of the trial: 12 months Expected start date: December 2019 Objectives: Principal:To verify the changes in plasma PPi, and the main molecules that regulate it (NPP1-3, TNAP) after oral administration of lansoprazole in patients diagnosed with PXE.

Description of treatment:

Selection:20 patients who meet all the criteria for inclusion and none for exclusion.

Randomisation and 1st stage: Patients will receive lansoprazole 30mg/day or their placebo for 8 weeks.

Wash-out: After 8 weeks, all treatment will be suspended for 15 days. 2nd stage (crossed): Treatment is crossed, each patient serves as his or her own control.

Evaluation variables:

1. Date of Birth
2. Sex.
3. Physical examination (anthropometry and vital signs)
4. Date of first symptom.
5. Date of final diagnosis
6. Ocular affectation (orange peel skin, complete striae angioides, lucentis, corrected visual acuity, cataracts, intraocular pressure, fundus (vascular flow, optic nerve drusen, retinal atrophy, neovascular membranes, macular thickness, colloid thickness).
7. Skin affectation (yellowish papules or plaques on the side of the neck or other areas of flexure and lax skin).
8. Vascular affectation (intermittent claudication clinic, angina and/or episode of acute myocardial infarction and/or non-embolic ischemic stroke, surgical or percutaneous revascularisation, cardiac murmur,10.)
9. History of renal lithiasis, arterial hypertension, diabetes mellitus, treatments, smoking and dyslipidemia.
10. Specific biochemical variables:

Inorganic pyrophosphate (IPP) NPP1 and NPP2.3: activity and mass concentration of the enzyme Non-specific tissue alkaline phosphatase (NTAP) and PHA. Osteocalcin: To check possible side effects on bone metabolism. 5'-Nucleotidas General analytical parameters (haemoglobin, haematocrit, MVC, MHC, platelets, neutrophils, prothrombin activity, TPTA, thrombin time, ferritin, PCR, glycaemia, urea, creatinine, cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, uric acid, calcium, phosphorus, alkaline phosphatase, PTH). By means of routine clinical laboratory techniques. Number of patients: TOTAL : 20 patients(Competitive recruitment)

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old
2. Patients diagnosed with PXE according to 2010 criteria by PLOMP et al.
3. At least, patients meet two of the following criteria:

   1. Retinal lesions such as Orange peel and/or Angioid streaks
   2. Skin lesions such as papules or yellowish plaques on the lateral face of the neck and / or flexures of the body (armpits, elbows, knees) or alterations in the skin biopsy with fragmentation and / or conglomerates of and / or calcification of the elastic fibers.
   3. A pathogenic mutation of the two alleles of the ABCC6 gene.

Exclusion Criteria:

1. Refusal of informed consent.
2. Vegetarian diet or extreme diets.
3. Pregnancy or its intention during the months of the study.
4. Age <18 years old
5. Known hypersensitivity to "prazoles" or proton pump inhibitors.
6. Intake of medications that may interfere with Lansoprazole and that cannot be withdrawn or modified in its form of administration to avoid such interference.
7. Prior taking of proton pump inhibitors, except for a wash out period of 15 days if the clinical situation of the patient allows it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-06-24 (Estimated); Study Completion 2021-06-24 (Estimated)

PRIMARY OUTCOMES:
Changes in PPi,NPP1-3 and TNAP | 8 weeks, 18 weeks
  changes in plasma PPi, and the main molecules that regulate it (NPP1-3, TNAP) after oral administration of lansoprazole in patients diagnosed with PXE

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain

REFERENCES:
- [Background] Le Saux O, Urban Z, Tschuch C, Csiszar K, Bacchelli B, Quaglino D, Pasquali-Ronchetti I, Pope FM, Richards A, Terry S, Bercovitch L, de Paepe A, Boyd CD. Mutations in a gene encoding an ABC transporter cause pseudoxanthoma elasticum. Nat Genet. 2000 Jun;25(2):223-7. doi: 10.1038/76102. PMID 10835642
- [Background] Scheffer GL, Hu X, Pijnenborg AC, Wijnholds J, Bergen AA, Scheper RJ. MRP6 (ABCC6) detection in normal human tissues and tumors. Lab Invest. 2002 Apr;82(4):515-8. doi: 10.1038/labinvest.3780444. No abstract available. PMID 11950908
- [Background] Brown SJ, Talks SJ, Needham SJ, Taylor AE. Pseudoxanthoma elasticum: biopsy of clinically normal skin in the investigation of patients with angioid streaks. Br J Dermatol. 2007 Oct;157(4):748-51. doi: 10.1111/j.1365-2133.2007.08076.x. Epub 2007 Jul 30. PMID 17666106
- [Background] Schroder F, Hausser I, Szliska C, Lawall H, Diehm C. Images in vascular medicine. Pseudoxanthoma elasticum: under-recognized cause of early onset peripheral arterial disease? Vasc Med. 2006 Nov;11(4):266-7. doi: 10.1177/1358863x06075186. No abstract available. PMID 17390553
- [Background] Fabre B, Bayle P, Bazex J, Durand D, Lamant L, Chassaing N. Pseudoxanthoma elasticum and nephrolithiasis. J Eur Acad Dermatol Venereol. 2005 Mar;19(2):212-5. doi: 10.1111/j.1468-3083.2005.01007.x. PMID 15752294
- [Background] Chassaing N, Martin L, Calvas P, Le Bert M, Hovnanian A. Pseudoxanthoma elasticum: a clinical, pathophysiological and genetic update including 11 novel ABCC6 mutations. J Med Genet. 2005 Dec;42(12):881-92. doi: 10.1136/jmg.2004.030171. Epub 2005 May 13. PMID 15894595
- [Background] Laube S, Moss C. Pseudoxanthoma elasticum. Arch Dis Child. 2005 Jul;90(7):754-6. doi: 10.1136/adc.2004.062075. PMID 15970621
- [Background] Li Q, Jiang Q, Pfendner E, Varadi A, Uitto J. Pseudoxanthoma elasticum: clinical phenotypes, molecular genetics and putative pathomechanisms. Exp Dermatol. 2009 Jan;18(1):1-11. doi: 10.1111/j.1600-0625.2008.00795.x. Epub 2008 Oct 22. PMID 19054062
- [Background] Lebwohl M, Schwartz E, Lemlich G, Lovelace O, Shaikh-Bahai F, Fleischmajer R. Abnormalities of connective tissue components in lesional and non-lesional tissue of patients with pseudoxanthoma elasticum. Arch Dermatol Res. 1993;285(3):121-6. doi: 10.1007/BF01112912. PMID 8503691
- [Background] Plomp AS, Toonstra J, Bergen AA, van Dijk MR, de Jong PT. Proposal for updating the pseudoxanthoma elasticum classification system and a review of the clinical findings. Am J Med Genet A. 2010 Apr;152A(4):1049-58. doi: 10.1002/ajmg.a.33329. PMID 20358627
- [Background] Quaglino D, Sartor L, Garbisa S, Boraldi F, Croce A, Passi A, De Luca G, Tiozzo R, Pasquali-Ronchetti I. Dermal fibroblasts from pseudoxanthoma elasticum patients have raised MMP-2 degradative potential. Biochim Biophys Acta. 2005 Jun 30;1741(1-2):42-7. doi: 10.1016/j.bbadis.2004.09.012. Epub 2004 Oct 8. PMID 15955448
- [Background] Pasquali-Ronchetti I, Garcia-Fernandez MI, Boraldi F, Quaglino D, Gheduzzi D, De Vincenzi Paolinelli C, Tiozzo R, Bergamini S, Ceccarelli D, Muscatello U. Oxidative stress in fibroblasts from patients with pseudoxanthoma elasticum: possible role in the pathogenesis of clinical manifestations. J Pathol. 2006 Jan;208(1):54-61. doi: 10.1002/path.1867. PMID 16261549
- [Background] Quaglino D, Boraldi F, Barbieri D, Croce A, Tiozzo R, Pasquali Ronchetti I. Abnormal phenotype of in vitro dermal fibroblasts from patients with Pseudoxanthoma elasticum (PXE). Biochim Biophys Acta. 2000 Apr 15;1501(1):51-62. doi: 10.1016/s0925-4439(00)00007-7. PMID 10727849
- [Background] Ronchetti I, Boraldi F, Annovi G, Cianciulli P, Quaglino D. Fibroblast involvement in soft connective tissue calcification. Front Genet. 2013 Mar 5;4:22. doi: 10.3389/fgene.2013.00022. eCollection 2013. PMID 23467434
- [Background] Boraldi F, Annovi G, Bartolomeo A, Quaglino D. Fibroblasts from patients affected by Pseudoxanthoma elasticum exhibit an altered PPi metabolism and are more responsive to pro-calcifying stimuli. J Dermatol Sci. 2014 Apr;74(1):72-80. doi: 10.1016/j.jdermsci.2013.12.008. Epub 2014 Jan 2. PMID 24461675
- [Background] Boraldi F, Bartolomeo A, Li Q, Uitto J, Quaglino D. Changes in dermal fibroblasts from Abcc6(-/-) mice are present before and after the onset of ectopic tissue mineralization. J Invest Dermatol. 2014 Jul;134(7):1855-1861. doi: 10.1038/jid.2014.88. Epub 2014 Feb 13. PMID 24670382
- [Background] Garcia-Fernandez MI, Gheduzzi D, Boraldi F, Paolinelli CD, Sanchez P, Valdivielso P, Morilla MJ, Quaglino D, Guerra D, Casolari S, Bercovitch L, Pasquali-Ronchetti I. Parameters of oxidative stress are present in the circulation of PXE patients. Biochim Biophys Acta. 2008 Jul-Aug;1782(7-8):474-81. doi: 10.1016/j.bbadis.2008.05.001. Epub 2008 May 10. PMID 18513494
- [Background] Morillo MJ, Mora J, Soler A, Garcia-Campos JM, Garcia-Fernandez I, Sanchez P, Valdivieso P. [Retinal autofluorescence imaging in patients with pseudoxanthoma elasticum]. Arch Soc Esp Oftalmol. 2011 Jan;86(1):8-15. doi: 10.1016/j.oftal.2010.11.019. Epub 2011 Feb 20. Spanish. PMID 21414524
- [Background] Jiang Q, Endo M, Dibra F, Wang K, Uitto J. Pseudoxanthoma elasticum is a metabolic disease. J Invest Dermatol. 2009 Feb;129(2):348-54. doi: 10.1038/jid.2008.212. Epub 2008 Aug 14. PMID 18685618
- [Background] Uitto J, Li Q, Jiang Q. Pseudoxanthoma elasticum: molecular genetics and putative pathomechanisms. J Invest Dermatol. 2010 Mar;130(3):661-70. doi: 10.1038/jid.2009.411. Epub 2009 Dec 24. PMID 20032990
- [Background] Boraldi F, Garcia-Fernandez M, Paolinelli-Devincenzi C, Annovi G, Schurgers L, Vermeer C, Cianciulli P, Ronchetti I, Quaglino D. Ectopic calcification in beta-thalassemia patients is associated with increased oxidative stress and lower MGP carboxylation. Biochim Biophys Acta. 2013 Dec;1832(12):2077-84. doi: 10.1016/j.bbadis.2013.07.017. Epub 2013 Jul 27. PMID 23899606
- [Background] Li Q, Jiang Q, Uitto J. Ectopic mineralization disorders of the extracellular matrix of connective tissue: molecular genetics and pathomechanisms of aberrant calcification. Matrix Biol. 2014 Jan;33:23-8. doi: 10.1016/j.matbio.2013.06.003. Epub 2013 Jul 25. PMID 23891698
- [Background] Jansen RS, Kucukosmanoglu A, de Haas M, Sapthu S, Otero JA, Hegman IE, Bergen AA, Gorgels TG, Borst P, van de Wetering K. ABCC6 prevents ectopic mineralization seen in pseudoxanthoma elasticum by inducing cellular nucleotide release. Proc Natl Acad Sci U S A. 2013 Dec 10;110(50):20206-11. doi: 10.1073/pnas.1319582110. Epub 2013 Nov 25. PMID 24277820
- [Background] Jansen RS, Duijst S, Mahakena S, Sommer D, Szeri F, Varadi A, Plomp A, Bergen AA, Oude Elferink RP, Borst P, van de Wetering K. ABCC6-mediated ATP secretion by the liver is the main source of the mineralization inhibitor inorganic pyrophosphate in the systemic circulation-brief report. Arterioscler Thromb Vasc Biol. 2014 Sep;34(9):1985-9. doi: 10.1161/ATVBAHA.114.304017. Epub 2014 Jun 26. PMID 24969777
- [Background] Moore SN, Tanner SB, Schoenecker JG. Bisphosphonates: from softening water to treating PXE. Cell Cycle. 2015;14(9):1354-5. doi: 10.1080/15384101.2015.1024585. No abstract available. PMID 25894689
- [Background] Narisawa S, Harmey D, Yadav MC, O'Neill WC, Hoylaerts MF, Millan JL. Novel inhibitors of alkaline phosphatase suppress vascular smooth muscle cell calcification. J Bone Miner Res. 2007 Nov;22(11):1700-10. doi: 10.1359/jbmr.070714. PMID 17638573
- [Background] Li Q, Sundberg JP, Levine MA, Terry SF, Uitto J. The effects of bisphosphonates on ectopic soft tissue mineralization caused by mutations in the ABCC6 gene. Cell Cycle. 2015;14(7):1082-9. doi: 10.1080/15384101.2015.1007809. PMID 25607347
- [Background] Millán JL (2006) APs as Physiological and Disease Markers. In Mammalian Alkaline Phosphatases, pp. 165-185: Wiley-VCH Verlag GmbH & Co. KgaA
- [Background] Boraldi F, Annovi G, Guerra D, Paolinelli Devincenzi C, Garcia-Fernandez MI, Panico F, De Santis G, Tiozzo R, Ronchetti I, Quaglino D. Fibroblast protein profile analysis highlights the role of oxidative stress and vitamin K recycling in the pathogenesis of pseudoxanthoma elasticum. Proteomics Clin Appl. 2009 Sep;3(9):1084-98. doi: 10.1002/prca.200900007. Epub 2009 Aug 26. PMID 21137008
- [Background] Boraldi F, Quaglino D, Croce MA, Garcia Fernandez MI, Tiozzo R, Gheduzzi D, Bacchelli B, Pasquali Ronchetti I. Multidrug resistance protein-6 (MRP6) in human dermal fibroblasts. Comparison between cells from normal subjects and from Pseudoxanthoma elasticum patients. Matrix Biol. 2003 Nov;22(6):491-500. doi: 10.1016/j.matbio.2003.09.001. PMID 14667841
- [Background] Delomenede M, Buchet R, Mebarek S. Lansoprazole is an uncompetitive inhibitor of tissue-nonspecific alkaline phosphatase. Acta Biochim Pol. 2009;56(2):301-5. Epub 2009 Jun 18. PMID 19543559
- [Background] Matsunaga C, Izumi S, Furukubo T, Satoh M, Yamakawa T, Uchida T, Kadowaki D, Hirata S. Effect of famotidine and lansoprazole on serum phosphorus levels in hemodialysis patients on calcium carbonate therapy. Clin Nephrol. 2007 Aug;68(2):93-8. doi: 10.5414/cnp68093. PMID 17722708
- [Background] O'Neill WC, Sigrist MK, McIntyre CW. Plasma pyrophosphate and vascular calcification in chronic kidney disease. Nephrol Dial Transplant. 2010 Jan;25(1):187-91. doi: 10.1093/ndt/gfp362. Epub 2009 Jul 24. PMID 19633093
- [Background] Battisti V, Maders LD, Bagatini MD, Battisti IE, Belle LP, Santos KF, Maldonado PA, Thome GR, Schetinger MR, Morsch VM. Ectonucleotide pyrophosphatase/phosphodiesterase (E-NPP) and adenosine deaminase (ADA) activities in prostate cancer patients: influence of Gleason score, treatment and bone metastasis. Biomed Pharmacother. 2013 Apr;67(3):203-8. doi: 10.1016/j.biopha.2012.12.004. Epub 2012 Dec 26. PMID 23433854
- [Background] Sergienko E, Su Y, Chan X, Brown B, Hurder A, Narisawa S, Millan JL. Identification and characterization of novel tissue-nonspecific alkaline phosphatase inhibitors with diverse modes of action. J Biomol Screen. 2009 Aug;14(7):824-37. doi: 10.1177/1087057109338517. Epub 2009 Jun 25. PMID 19556612